CLINICAL TRIAL: NCT03749226
Title: Efficacy, Safety and Pharmacokinetics Profile of Nebulized Aztreonam Lysine (AZLI) for Prevention of Gram Negative Pneumonia in Heavily Colonized Mechanically Ventilated Patients
Brief Title: Nebulized Aztreonam for Prevention of Gram Negative Ventilator-associated Pneumonia
Acronym: AZLIS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: due to COVID-19 pandemia
Sponsor: Hospital Universitari Joan XXIII de Tarragona. (Other)
Responsible Party: Principal Investigator, Alejandro Rodriguez Oviedo , MD, Principal Investigator, Hospital Universitari Joan XXIII de Tarragona.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AZLI-2018-AR
Record Dates: First submitted 2018-04-20; First posted 2018-11-21 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Ventilator Associated Pneumonia; Prevention; Respiratory Infection Other
Keywords: Nebulized antibiotic; Ventilator associated pneumonia; Ventilated associated tracheobronchitis; Aztreonam lysine
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: Twenty consecutive patients heavily colonized by Gram-negative bacteria will be eligible for this study. Patients will be randomized to receive either AZLI nebulized or nothing via 1:1 randomization at study or control group.
  Patients assigned to study group will receive nebulized Aztreonam lysine (AZLI 75 mg-dose) three times /day during 5 days by mean of the ultrasonic nebulizer (Aeroneb solo®) plus Combihaler® spacer adapted of the ventilator. All patients will be on conventional volume-control ventilator setting during the antibiotic therapy. Systemic antibiotics will not be used in any patient. If the attending physician saw the need to administer intravenous antibiotics after the patient has entry in the study, this patients should be removed from the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZLI group (Active Comparator): Patients assigned to study group will receive nebulized Aztreonam lysine (AZLI 75 mg-dose) three times /day during 5 days by mean of the ultrasonic nebulizer (Aeroneb solo®) plus Combihaler® spacer adapted of the ventilator
  Interventions: Drug: Aztreonam lysine; Device: Aerogen Solo; Device: CombiHaler
- Control group (No Intervention): Patients assigned to control group will no receive any intervention for heavy Gram negative colonization

INTERVENTIONS:
Drug: Aztreonam lysine — nebulization
  Arms: AZLI group
Device: Aerogen Solo — Aerogen's vibrating mesh technology, available within the Aerogen® Solo has been adopted for use of conventional mechanical ventilation. Aerogen Solo utilizes active vibrating mesh technology, where energy applied to the vibrational element, causes vibration of each of the 1000 funnel shaped apertures within the mesh. The mesh acts as a micropump drawing liquid through the holes producing a low velocity aerosol optimized for targeted drug delivery to the lungs. According our study (Rodriguez A et al , Expert Opin Drug Deliv. 2017 Dec;14(12):1447-1453) Aeroneb Solo showed an excellent aerosol delivery profile for Aztreonam lysine (AZLI) in an in vitro model of MV with short drug delivery time.
  Arms: AZLI group
Device: CombiHaler — The inhalation chamber CombiHaler™ spacer for mechanical ventilation and critical care (ICU) allows using both a vibrating mesh nebulizer such as Aeroneb ™, and a pMDI. It saves 50% of the nebulized drug when used in invasive ventilation. The inhalation chamber CombiHaler® is integrated on a circuit of a breathing device in invasive ventilation in particular for connexion of an Aeroneb® Pro or an Aeroneb® Solo. According our study (Rodriguez A et al , Expert Opin Drug Deliv. 2017 Dec;14(12):1447-1453) a better aerosol delivery performance (30%) was obtained using the Conbihaler spacer.
  Arms: AZLI group

SUMMARY:
Aerosol antibiotic administration offers the theoretical advantages of achieving high drug concentration at the infection site and low systemic absorption, thereby avoiding toxicity. Antibiotic aerosolization has good results in patients with cystic fibrosis, but data are scarce for patients under mechanical ventilation.

Prospective, randomized 1:1, open-label study to assess the microbiological cure and pharmacokinetics (PK), safety and efficacy of nebulized Aztreonam lysine (75 mg dose) each 8 hr during 5 days in ventilated patients heavily colonized by Gram-negative bacteria. It is planned to include a total of 20 ventilated patients heavily colonized. Only ten of them (active group) will receive 5 days of treatment with nebulized AZLI.The control group will not receive treatment.

DETAILED DESCRIPTION:
The main objectives of this study is:

To compare the microbiological cure at day 5 of treatment and the incidence of Gram-negative IVAC between 7th and 10th days after last dose in patients heavily colonized by Gram-negative bacteria treated with nebulized AZLI vs. no treatment.

The secundary objective of this study are:

1. Safety and tolerability of AZLI administered during 5 days in adults patients under mechanical ventilation heavily colonized by Gram-negative bacteria
2. The pharmacokinetic profile in endotracheal aspirate (EA) or bronchoalveolar lavage (BAL).
3. The plasma levels of nebulized AZLI in patients under mechanical ventilation heavily colonized by Gram-negative bacteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patients under mechanical ventilation for more than 5 day.
3. Patient with heavy colonization by Gram-negative microorganisms.
4. No clinical suspicion of infections-related ventilator-associated complications (IVAC) according CDC criteria (Figure 1).
5. Patients or his/her legal representative with ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and to return for the required assessments.
6. Informed consent signed

Exclusion Criteria:

1. Suspected of IVAC.
2. Patients with known hypersensitivity to Aztreonam.
3. Patients who received more than 48 hours of broad spectrum antibiotics.
4. Evidence of active mycobacterium infections, chronic pulmonary infection or bronchial obstruction.
5. Granulomatous disease, lung cancer or lung transplant.
6. Acute respiratory distress syndrome (ARDS)
7. Woman who is pregnant or breast-feeding while enrolled in this study.
8. Any medical condition which, in the opinion of the Investigator, places the patient at an unacceptable risk for toxicities if entered into the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Microbiological cure | 5 days
  Microbiological cure was defined as endotracheal aspirate (EA) or BAL cultures with consistently negative results after five day of therapy.

SECONDARY OUTCOMES:
Pharmacokinetic of aztreonam lysine in respiratory samples | day 0 and day 2
  Maximum bronchial concentration[Cmax]
Pharmacokinetic of aztreonam lysine in respiratory samples | day 0 and day 2
  time to maximum bronchial concentration[Tmax]
Pharmacokinetic of aztreonam lysine in respiratory samples | day 0 and day 2
  Maximum bronchial concentration [Cmax] in tracheal aspirate (EA) or bronchoalveolar lavage (BAL) samples
Pharmacokinetic of aztreonam lysine in respiratory samples | day 0 and day 2
  Area under the bronchial concentration-time curve [AUC] in tracheal aspirate (EA) or bronchoalveolar lavage (BAL) samples
Pharmacokinetic of aztreonam lysine in respiratory samples | day 0 and day 2
  Terminal elimination half-time [t1/2] in tracheal aspirate (EA) or bronchoalveolar lavage (BAL) samples
Pharmacokinetic profile of aztreonam lysine in serum samples | day 3
  Time to maximum serum concentration[Tmax] in serum samples
Pharmacokinetic profile of aztreonam lysine in serum samples | day 3
  Area under the serum concentration-time curve [AUC] in serum samples
Pharmacokinetic profile of aztreonam lysine in serum samples | day 3
  Terminal elimination half-time [t1/2] in serum samples
SAEs and AEs assessments | 10 days
  adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Critical Care Department - Hospital Universitario de Tarragona Joan XXIII, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klompas M. Ventilator-associated events surveillance: a patient safety opportunity. Curr Opin Crit Care. 2013 Oct;19(5):424-31. doi: 10.1097/MCC.0b013e3283636bc9. PMID 23778075
- [Background] File TM Jr. New diagnostic tests for pneumonia: what is their role in clinical practice? Clin Chest Med. 2011 Sep;32(3):417-30. doi: 10.1016/j.ccm.2011.05.011. Epub 2011 Jul 12. PMID 21867812
- [Background] Niederman MS. Respiratory tract infections: advances in diagnosis, management and prevention. Clin Chest Med. 2011 Sep;32(3):xiii-xiv. doi: 10.1016/j.ccm.2011.07.001. No abstract available. PMID 21867811
- [Background] Craven DE. Ventilator-associated tracheobronchitis (VAT): questions, answers, and a new paradigm? Crit Care. 2008;12(3):157. doi: 10.1186/cc6912. Epub 2008 Jun 18. PMID 18598373
- [Background] Craven DE, Chroneou A, Zias N, Hjalmarson KI. Ventilator-associated tracheobronchitis: the impact of targeted antibiotic therapy on patient outcomes. Chest. 2009 Feb;135(2):521-528. doi: 10.1378/chest.08-1617. Epub 2008 Sep 23. PMID 18812452
- [Background] Nseir S, Ader F, Marquette CH. Nosocomial tracheobronchitis. Curr Opin Infect Dis. 2009 Apr;22(2):148-53. doi: 10.1097/QCO.0b013e3283229fdb. PMID 19276882
- [Background] Chastre J, Fagon JY. Ventilator-associated pneumonia. Am J Respir Crit Care Med. 2002 Apr 1;165(7):867-903. doi: 10.1164/ajrccm.165.7.2105078. PMID 11934711
- [Background] Nseir S, Di Pompeo C, Pronnier P, Beague S, Onimus T, Saulnier F, Grandbastien B, Mathieu D, Delvallez-Roussel M, Durocher A. Nosocomial tracheobronchitis in mechanically ventilated patients: incidence, aetiology and outcome. Eur Respir J. 2002 Dec;20(6):1483-9. doi: 10.1183/09031936.02.00012902. PMID 12503708
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Kollef MH, Hamilton CW, Montgomery AB. Aerosolized antibiotics: do they add to the treatment of pneumonia? Curr Opin Infect Dis. 2013 Dec;26(6):538-44. doi: 10.1097/QCO.0000000000000004. PMID 24126716
- [Background] Venier AG, Leroyer C, Slekovec C, Talon D, Bertrand X, Parer S, Alfandari S, Guerin JM, Megarbane B, Lawrence C, Clair B, Lepape A, Perraud M, Cassier P, Trivier D, Boyer A, Dubois V, Asselineau J, Rogues AM, Thiebaut R; DYNAPYO study group. Risk factors for Pseudomonas aeruginosa acquisition in intensive care units: a prospective multicentre study. J Hosp Infect. 2014 Oct;88(2):103-8. doi: 10.1016/j.jhin.2014.06.018. Epub 2014 Aug 1. PMID 25155240
- [Background] Drakulovic MB, Bauer TT, Torres A, Gonzalez J, Rodriguez MJ, Angrill J. Initial bacterial colonization in patients admitted to a respiratory intensive care unit: bacteriological pattern and risk factors. Respiration. 2001;68(1):58-66. doi: 10.1159/000050464. PMID 11223732
- [Background] Azim A, Dwivedi M, Rao PB, Baronia AK, Singh RK, Prasad KN, Poddar B, Mishra A, Gurjar M, Dhole TN. Epidemiology of bacterial colonization at intensive care unit admission with emphasis on extended-spectrum beta-lactamase- and metallo-beta-lactamase-producing Gram-negative bacteria--an Indian experience. J Med Microbiol. 2010 Aug;59(Pt 8):955-960. doi: 10.1099/jmm.0.018085-0. Epub 2010 Apr 22. PMID 20413621
- [Background] Horianopoulou M, Legakis NJ, Kanellopoulou M, Lambropoulos S, Tsakris A, Falagas ME. Frequency and predictors of colonization of the respiratory tract by VIM-2-producing Pseudomonas aeruginosa in patients of a newly established intensive care unit. J Med Microbiol. 2006 Oct;55(Pt 10):1435-1439. doi: 10.1099/jmm.0.46713-0. PMID 17005794
- [Background] Ramsey BW, Pepe MS, Quan JM, Otto KL, Montgomery AB, Williams-Warren J, Vasiljev-K M, Borowitz D, Bowman CM, Marshall BC, Marshall S, Smith AL. Intermittent administration of inhaled tobramycin in patients with cystic fibrosis. Cystic Fibrosis Inhaled Tobramycin Study Group. N Engl J Med. 1999 Jan 7;340(1):23-30. doi: 10.1056/NEJM199901073400104. PMID 9878641
- [Background] Assael BM, Pressler T, Bilton D, Fayon M, Fischer R, Chiron R, LaRosa M, Knoop C, McElvaney N, Lewis SA, Bresnik M, Montgomery AB, Oermann CM; AZLI Active Comparator Study Group. Inhaled aztreonam lysine vs. inhaled tobramycin in cystic fibrosis: a comparative efficacy trial. J Cyst Fibros. 2013 Mar;12(2):130-40. doi: 10.1016/j.jcf.2012.07.006. Epub 2012 Sep 15. PMID 22985692
- [Background] Coates AL, Green M, Leung K, Chan J, Ribeiro N, Louca E, Ratjen F, Charron M, Tservistas M, Keller M. Rapid pulmonary delivery of inhaled tobramycin for Pseudomonas infection in cystic fibrosis: a pilot project. Pediatr Pulmonol. 2008 Aug;43(8):753-9. doi: 10.1002/ppul.20850. PMID 18613006
- [Background] Gibson RL, Retsch-Bogart GZ, Oermann C, Milla C, Pilewski J, Daines C, Ahrens R, Leon K, Cohen M, McNamara S, Callahan TL, Markus R, Burns JL. Microbiology, safety, and pharmacokinetics of aztreonam lysinate for inhalation in patients with cystic fibrosis. Pediatr Pulmonol. 2006 Jul;41(7):656-65. doi: 10.1002/ppul.20429. PMID 16703579
- [Background] Poulakou G, Siakallis G, Tsiodras S, Arfaras-Melainis A, Dimopoulos G. Nebulized antibiotics in mechanically ventilated patients: roadmap and challenges. Expert Rev Anti Infect Ther. 2017 Mar;15(3):211-229. doi: 10.1080/14787210.2017.1268052. Epub 2017 Jan 2. PMID 27921442
- [Background] Kalil AC, Metersky ML, Klompas M, Muscedere J, Sweeney DA, Palmer LB, Napolitano LM, O'Grady NP, Bartlett JG, Carratala J, El Solh AA, Ewig S, Fey PD, File TM Jr, Restrepo MI, Roberts JA, Waterer GW, Cruse P, Knight SL, Brozek JL. Management of Adults With Hospital-acquired and Ventilator-associated Pneumonia: 2016 Clinical Practice Guidelines by the Infectious Diseases Society of America and the American Thoracic Society. Clin Infect Dis. 2016 Sep 1;63(5):e61-e111. doi: 10.1093/cid/ciw353. Epub 2016 Jul 14. PMID 27418577
- [Background] Palmer LB. Ventilator-associated infection: the role for inhaled antibiotics. Curr Opin Pulm Med. 2015 May;21(3):239-49. doi: 10.1097/MCP.0000000000000160. PMID 25784247
- [Background] Rodriguez A, Barcenilla F. Nebulized antibiotics. An adequate option for treating ventilator-associated respiratory infection? Med Intensiva. 2015 Mar;39(2):97-100. doi: 10.1016/j.medin.2014.10.006. Epub 2015 Feb 2. English, Spanish. PMID 25655673
- [Background] Dugernier J, Wittebole X, Roeseler J, Michotte JB, Sottiaux T, Dugernier T, Laterre PF, Reychler G. Influence of inspiratory flow pattern and nebulizer position on aerosol delivery with a vibrating-mesh nebulizer during invasive mechanical ventilation: an in vitro analysis. J Aerosol Med Pulm Drug Deliv. 2015 Jun;28(3):229-36. doi: 10.1089/jamp.2014.1131. Epub 2014 Nov 13. PMID 25393556
- [Background] Oermann CM, McCoy KS, Retsch-Bogart GZ, Gibson RL, McKevitt M, Montgomery AB. Pseudomonas aeruginosa antibiotic susceptibility during long-term use of aztreonam for inhalation solution (AZLI). J Antimicrob Chemother. 2011 Oct;66(10):2398-404. doi: 10.1093/jac/dkr303. Epub 2011 Jul 22. PMID 21784781
- [Background] McCoy KS, Quittner AL, Oermann CM, Gibson RL, Retsch-Bogart GZ, Montgomery AB. Inhaled aztreonam lysine for chronic airway Pseudomonas aeruginosa in cystic fibrosis. Am J Respir Crit Care Med. 2008 Nov 1;178(9):921-8. doi: 10.1164/rccm.200712-1804OC. Epub 2008 Jul 24. PMID 18658109
- [Result] Martin-Loeches I, Povoa P, Rodriguez A, Curcio D, Suarez D, Mira JP, Cordero ML, Lepecq R, Girault C, Candeias C, Seguin P, Paulino C, Messika J, Castro AG, Valles J, Coelho L, Rabello L, Lisboa T, Collins D, Torres A, Salluh J, Nseir S; TAVeM study. Incidence and prognosis of ventilator-associated tracheobronchitis (TAVeM): a multicentre, prospective, observational study. Lancet Respir Med. 2015 Nov;3(11):859-68. doi: 10.1016/S2213-2600(15)00326-4. Epub 2015 Oct 22. PMID 26472037
- [Result] Nseir S, Povoa P, Salluh J, Rodriguez A, Martin-Loeches I. Is there a continuum between ventilator-associated tracheobronchitis and ventilator-associated pneumonia? Intensive Care Med. 2016 Jul;42(7):1190-2. doi: 10.1007/s00134-016-4283-x. Epub 2016 Apr 14. No abstract available. PMID 27080532
- [Result] Boukhettala N, Poree T, Diot P, Vecellio L. In vitro performance of spacers for aerosol delivery during adult mechanical ventilation. J Aerosol Med Pulm Drug Deliv. 2015 Apr;28(2):130-6. doi: 10.1089/jamp.2013.1091. Epub 2014 Jul 22. PMID 25050644
- [Result] McKindley DS, Boucher BA, Hess MM, Croce MA, Fabian TC. Pharmacokinetics of aztreonam and imipenem in critically ill patients with pneumonia. Pharmacotherapy. 1996 Sep-Oct;16(5):924-31. PMID 8888088
- [Result] Rodriguez A, Cabrera M, Reyes LF, Bodi M, Trefler S, Canadell L, Barahona D, Ehrmann S, Martin-Loeches I, Restrepo MI, Vecellio L. In vitro evaluation of aerosol delivery of aztreonam lysine (AZLI): an adult mechanical ventilation model. Expert Opin Drug Deliv. 2017 Dec;14(12):1447-1453. doi: 10.1080/17425247.2017.1393411. Epub 2017 Oct 23. PMID 29041861